CLINICAL TRIAL: NCT05708196
Title: Evaluation of β-tricalcium Phosphate/Calcium Sulfate Versus Allografts in Implant Bone Reconstructive Procedures; A Histological and Radiographical Clinical Trial.
Brief Title: Evaluation of β-tricalcium Phosphate/Calcium Sulfate Versus Allografts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Heba Elsheikh, assistant professor of oral and maxillofacial surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M23011122
Record Dates: First submitted 2023-01-11; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Tooth Extraction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): ten extraction sockets left for normal healing (blood clot).
- group 2 (Experimental): ten extraction sockets filled with Alloplast bone grafting material (EthOss, Ethoss Regeneration Ltd, Silsden, UK).
  Interventions: Other: Alloplast bone grafting material (EthOss, Ethoss Regeneration Ltd, Silsden, UK).
- group 3 (Experimental): ten extraction sockets filled with Allograft bone grafting material.
  Interventions: Other: Allograft bone grafting material.

INTERVENTIONS:
Other: Alloplast bone grafting material (EthOss, Ethoss Regeneration Ltd, Silsden, UK). — After tooth extraction, the tooth socket will begrafted with Alloplast grafting material
  Arms: group 2
Other: Allograft bone grafting material. — After tooth extraction, the tooth socket will be grafted with allograft grafting material
  Arms: group 3

SUMMARY:
Thirty healthy patients will be selected from the outpatient clinic of the Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Mansoura University, to be included in this study with non-restorable posterior teeth.Patients will be selected according to the following criteria: 1) having a non-restorable posterior tooth. 2) being healthy, with no systemic diseases that might contraindicate receiving a dental implant. 3) having good oral hygiene. 4) aged between 18 to 45 years old. 5) having sufficient alveolar bone volume and height at the future implant site.Patients were classified into three groups:

* Group I: ten extraction sockets left for normal healing (blood clot).
* Group II: ten extraction sockets filled with Alloplast bone grafting material (EthOss, Ethoss Regeneration Ltd, Silsden, UK).
* Group III: ten extraction sockets filled with Allograft bone grafting material.Evaluation and Follow-up

All patients will be evaluated clinically and radiographically during a follow up period of 4 months, where the following criteria will be evaluated:

A- Clinical evaluation:

* Patients will be evaluated at 1 week, 4 weeks and 8 weeks.
* Clinical evaluations of soft tissue healing, and keratinized tissue replacement will be assessed on the basis of the healing index proposed by Landry et al12.
* The scores will assess healing on the basis of redness, presence of granulation tissue, bleeding, suppuration, and epithelization.
* The surgical region will be examined clinically, if there is pain, redness, tissue resorption and bone graft stability.

B- Radiographic evaluation:

* Cone Beam Computed Tomography scan will be taken immediately after implant placement, and after 12 months.
* All patient scans will be taken by a Planmeca ProMax 3D unit (Planmeca OY, Helsinki, Finland) using fixed imaging parameter at every scan. All DICOM data will then be analyzed using On Demand 3D software (Version 1, Cyber Med, Seoul, South Korea).
* The vertical and horizontal measurements will be measured.
* The apico-coronal dimension will be calculated, the bottom of the socket will be considered the most apical point, whereas the alveolar bone margin will be considered the most coronal point of the socket bone wall.

C- Histological evaluation:

- Bone samples will be collected with trephine bur before implant placement, then fixed in 10% neutral buffered formalin for 24 hours, then transferred to 14% neutral buffered Ethylenediaminetetraacetic acid (EDTA) for decalcification 13. After confirming adequate decalcification, the specimens will be processed and embedded in paraffin blocks in the Pathology department, faculty of Medicine, Mansoura university for histological assessment, then stained with haematoxylin and eosin (H&E) as a routine stain to evaluate the quality of newly formed bone.

ELIGIBILITY:
Inclusion Criteria:

* having a non-restorable posterior tooth.
* being healthy, with no systemic diseases that might contraindicate receiving a dental implant.
* having good oral hygiene.
* aged between 18 to 45 years old.
* having sufficient alveolar bone volume and height at the future implant site

Exclusion Criteria:

* having received radiation therapy at the head and neck area or chemotherapy in the past 12 months.
* having uncontrolled diabetes.
* having poor oral hygiene or motivation.
* having bruxism or other parafunctional habit.
* having infection or inflammation at the proposed implant site.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Bone density measurement | 4 months
  CBCT will be used to assess bone density categories and HU

CONTACTS AND LOCATIONS:
Locations (1):
- Heba Elsheikh, Al Mansurah, Egypt